CLINICAL TRIAL: NCT02963740
Title: Feasibility of High Levels of Energy Expenditure From Physical Activity During a Weight Loss Intervention for Breast Cancer Survivors
Brief Title: Feasibility of High Levels of Energy Expenditure From Physical Activity for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004575
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer Female
Keywords: breast cancer survivor; weight loss program
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Loss Intervention Group (Experimental): Participants will take part in supervised exercise and home-based exercise sessions. Participants will be asked to follow a specific diet. Participants will be asked to take part in weekly behavioral group phone calls.
  Interventions: Behavioral: Supervised Exercise; Behavioral: Home-based Exercise; Behavioral: Group Phone Calls; Behavioral: Diet

INTERVENTIONS:
Behavioral: Supervised Exercise — Participants will take part in supervised exercise activities two times per week at a YMCA. Length of the activity will be increased during participation in study. Participants will start at 40 minutes per week and work their way up to 120 minutes per week.
Behavioral: Home-based Exercise — Aerobic exercise activities to be completed at home. Participants will be asked to start out doing 60 minutes at home and work up to 180 minutes of purposeful aerobic home exercise per week.
Behavioral: Group Phone Calls — Once weekly phone calls that are group-based. The calls will discuss lifestyle changes specific to participants and cover the effects of diet, physical activity, and weight on breast cancer risk, as well as body image and emotional eating.
Behavioral: Diet — Participants will consume a nutritionally balanced, reduced calorie diet as recommended by the Academy of Nutrition and Dietetics.

SUMMARY:
The purpose of the study is to demonstrate that breast cancer survivors who need to lose weight are able to follow a weight loss program which combines modest calorie restriction with a graduated activity program..

DETAILED DESCRIPTION:
Feasibility will be assessed by 1) the number of women that complete the 3--month program; 2) the number of women that can achieve the targeted amount of physical activity per week by the end of the program; and 3) the median amount of physical activity achieved group by all subjects that complete the program.

ELIGIBILITY:
Inclusion Criteria:

* Women < age 71 in good general health.
* Prior diagnosis of breast cancer.
* At least 3 months from completion of any cytotoxic chemotherapy or radiation or surgery. May continue to take endocrine therapy and/or maintenance trastuzumab.
* Body Mass Index (BMI) 30-45 kg/m2.
* By self-assessment, currently performing 60 minutes or less of purposeful exercise per week but able to walk at least 30 minutes on a level surface.
* Access to a smart phone capable of running MyFitnessPal and Garmin Connect apps and willing to have diet and exercise data from these apps viewed by study personnel.
* Live in the greater Kansas City Metropolitan Area
* Willing and able to perform moderate intensity exercise at least 5 days per week for 3 months.
* Willing to perform unsupervised home exercise for the entire 3 months.
* Willing to participate in a weekly behavioral modification group phone call for 3 months.
* Willing to participate in a controlled dietary intervention with portion controlled meals and partial meal and track food intake and exercise.

Exclusion Criteria:

* Use of metformin, insulin, steroids or weight loss or anti-psychotic drugs within the prior 3 weeks
* Individuals with prior bariatric surgery procedures
* Need for chronic immunosuppressive drugs
* Participation within the past 6 months on a structured weight loss program such as Weight Watchers®
* Physical impairments (bad hip, knees, feet, peripheral neuropathy) that would prohibit performing moderate intensity exercise at least 5 days per week.
* Any other condition or intercurrent illness that in the opinion of the investigator makes the subject a poor candidate for participation in the trial such as recent cardiac event.
* Currently receiving investigational agents in a clinical trial.

Max Age: 71 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Adherence to supervised exercise sessions | Week 12
  Adherence is defined as the percent of monitored sessions at the YMCA attended by the participant.

SECONDARY OUTCOMES:
Percent participants meeting physical activity goal | Week 9 to Week 12
  Measured as percentage of participants meeting final physical activity goal between week 9 to week 12. Measurement based off activity tracker participants will wear.
Compliance with group telephone sessions | Week 12
  Defined as number of participants attending at least 75% of the weekly group calls.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fabian CJ, Klemp JR, Marchello NJ, Vidoni ED, Sullivan DK, Nydegger JL, Phillips TA, Kreutzjans AL, Hendry B, Befort CA, Nye L, Powers KR, Hursting SD, Giles ED, Hamilton-Reeves JM, Li B, Kimler BF. Rapid Escalation of High-Volume Exercise during Caloric Restriction; Change in Visceral Adipose Tissue and Adipocytokines in Obese Sedentary Breast Cancer Survivors. Cancers (Basel). 2021 Sep 28;13(19):4871. doi: 10.3390/cancers13194871. PMID 34638355